CLINICAL TRIAL: NCT00283556
Title: Phase I/II Study of High Dose Irinotecan (Camptosar, CPT-11) in Patients With Recurrent Unresectable Malignant Glioma on Steroids/Anti-epileptics
Brief Title: High Dose Camptothecin-11 (CPT-11) in Recurrent Unresectable Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kentuckiana Cancer Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1068114; 44OE-ONC-0020-3
Record Dates: First submitted 2006-01-26; First posted 2006-01-30 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Malignant Glioma
Keywords: High Dose Irinotecan; CPT-11; Camptosar; Malignant Glioma; Unresectable
MeSH Terms: conditions — Glioma | interventions — Irinotecan

ARMS (3):
- Cohort #1 (Experimental): Cohort #1--Irinotecan 750 mg/m2 IV over 90 minutes every (Q) 3 weeks x 15 patients.
  Additional increments of 50 mg/m2 for subsequent cohorts until MTD is reached.
  Interventions: Drug: Irinotecan (Camptosar, CPT-11)
- Cohort #2 (Experimental): Cohort #2--Irinotecan 500 mg/m2 IV over 90 minutes Q 2 weeks x 3 patients.
  Additional increments of 50 mg/m2 for subsequent cohorts until MTD is reached.
  Interventions: Drug: Irinotecan (Camptosar, CPT-11)
- Cohort #3 (Experimental): Cohort #3--Irinotecan 600 mg/m2 IV over 90 minutes Q 2 weeks x 3 patients.
  Additional increments of 50 mg/m2 for subsequent cohorts until MTD is reached.
  Interventions: Drug: Irinotecan (Camptosar, CPT-11)

INTERVENTIONS:
Drug: Irinotecan (Camptosar, CPT-11) — Cohort #1--Irinotecan 750 mg/m2 IV over 90 minutes Q 3 weeks x 15 patients; Cohort #2--Irinotecan 500 mg/m2 IV over 90 minutes Q 2 weeks x 3 patients; Cohort #3--Irinotecan 600 mg/m2 IV over 90 minutes Q 2 weeks x 3 patients.
  Additional increments of 50 mg/m2 for subsequent cohorts until MTD is reached.

SUMMARY:
The purpose of this study is to compare the response to treatment and side effects associated with high dose irinotecan in patients with recurrent brain tumors.

DETAILED DESCRIPTION:
This is a phase I/II study of high dose irinotecan in patients with recurrent unresectable malignant glioma on steroids/anti-epileptics. The purpose is to compare the response to treatment and side effects associated with high dose irinotecan in patients with recurrent brain tumors.

ELIGIBILITY:
Inclusion Criteria:

* recurrent, unresectable primary CNS neoplasm per MRI
* ECOG status of 2 or less
* no prior therapy with camptothecans
* on an enzyme-inducing antiepileptic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to compare the response to treatment and side effects associated with high dose irinotecan in patients with recurrent brain tumors. | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Renato V. LaRocca, MD, Principal Investigator — Director
Locations (1):
- Kentuckiana Cancer Institute, Louisville, Kentucky, United States